CLINICAL TRIAL: NCT04928326
Title: Comparison of the InCardia Venous Pressure Diagnostic Technology CorWatch With Swan Ganz Catheter Measurements in the Cardiac Catheterization Laboratory and Cardiac Intensive Care Unit
Brief Title: Comparison of CorWatch With Right Heart Catheter Measurements in Heart Failure
Status: Completed | Type: Observational
Sponsor: InCardia Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CP-001A
Record Dates: First submitted 2021-06-08; First posted 2021-06-16 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure
Keywords: central venous pressure; right heart catheterization; hemodynamic congestion
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with heart failure undergoing right heart catheterization: Subjects with a diagnosis of NYHA class II-IV heart failure who meet the inclusion and exclusion criteria will be eligible for participation in this study.
  Interventions: Diagnostic Test: CorWatch

INTERVENTIONS:
Diagnostic Test: CorWatch — Non-invasive wearable monitor for the assessment of central venous pressure

SUMMARY:
This is an observational study to evaluate the agreement between the InCardia diagnostic technology CorWatch for the assessment of venous pressure in human subjects. This includes evaluation of InCardia technology in heart failure (HF) patients undergoing invasive right heart catheterization in a cardiac catheterization laboratory (cath lab) and in a cardiac intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with NYHA class II-IV heart failure irrespective of ejection fraction
* Patient is able to give consent

Exclusion Criteria:

* Severe tricuspid regurgitation
* Mechanical ventilation
* Patient is pregnant
* Inability to access either of the patient's upper arms.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of NYHA class II-IV heart failure who meet the inclusion and exclusion criteria will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Agreement with right atrial pressure as measured by Swan Ganz catheter | During the right heart catheterization procedure
  Agreement between the CVP/RAP as assessed by the CorWatchTM method and the right arterial pressure (RAP) as measured by SG catheter

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No